CLINICAL TRIAL: NCT04982276
Title: A Multicentre, Phase Ib/II Clinical Study of AK109 and AK104 With or Without Chemotherapy in Second-line Treatment of Advanced Gastric Adenocarcinoma or Gastroesophageal Junction Adenocarcinoma
Brief Title: A Study of AK109 and AK104 in Advanced Gastric Adenocarcinoma or Gastroesophageal Junction Adenocarcinoma
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Akeso (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: AK109-201
Record Dates: First submitted 2021-07-21; First posted 2021-07-29 (Actual); Last update posted 2025-11-19 (Actual); Status verified 2025-11

CONDITIONS: Gastric Adenocarcinoma and Gastroesophageal Junction Adenocarcinoma
MeSH Terms: interventions — Paclitaxel

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- AK109 combined with chemotherapy (Experimental): AK109 combined with paclitaxel, iv, every 3 weeks
  Interventions: Biological: AK109; Drug: paclitaxel
- AK104 and AK109 combined with chemotherapy (Experimental): AK104 combined with AK109 and paclitaxel, iv, every 3 weeks
  Interventions: Biological: AK109; Drug: paclitaxel; Biological: AK104

INTERVENTIONS:
Biological: AK109 — Subjects will receive AK109 by intravenous administration.
Drug: paclitaxel — Subjects will receive AK109 in combination with paclitaxel.
  Arms: AK109 combined with chemotherapy
Drug: paclitaxel — Subjects will receive AK104 and AK109 in combination with paclitaxel.
  Arms: AK104 and AK109 combined with chemotherapy
Biological: AK104 — Subjects will receive AK104 by intravenous administration.
  Arms: AK104 and AK109 combined with chemotherapy

SUMMARY:
This is a multicentre, Phase Ib/II Clinical Study of AK109 and AK104 With or Without Chemotherapy in Second-line Treatment of Advanced Gastric Adenocarcinoma or Gastroesophageal Junction Adenocarcinoma .

ELIGIBILITY:
Inclusion Criteria:

1. Written and signed informed consent
2. Age ≥ 18 years but ≤ 75 years
3. ECOG of 0 or 1.
4. Estimated life expectancy of ≥3 months.
5. Histologically or cytologically documented advanced unresectable or metastatic gastric adenocarcinoma or gastroesophageal Junction (GEJ) adenocarcinoma.
6. At least one measurable lesion per RECIST v1.1.
7. Gastric adenocarcinoma or gastroesophageal junction (GEJ) adenocarcinoma with failure of first-line treatment with anti-PD-1/L1 and chemotherapy
8. Adequate organ function.
9. Have agreed to take effective contraception from the date of signing the informed consent form until 120 days after the last administration.

Exclusion Criteria:

1. Other invasive malignancies within 3 years, except for locally treatable (manifested as cured) malignancies, such as basal or skin squamous cell carcinoma, superficial bladder cancer, cervical or breast carcinoma in situ.
2. Any previous systemic therapy targeting VEGF or anti-VEGFR signaling pathways.
3. In addition to PD1 or PD-L1,Prior exposure to anti-CTLA-4 antibody, or any other antibody or drug therapy for T cell co-stimulatory or checkpoint pathways, such as ICOS or agonists (e.g. CD40, CD137, GITR and OX40 etc).
4. Known history of primary immunodeficiency virus infection.
5. Known history of allogeneic organ transplantation or allogeneic hematopoietic stem cell transplantation.
6. Known history of interstitial lung disease.
7. Known history of active tuberculosis (TB).
8. Central nervous system (CNS) metastasis, meningeal metastasis, spinal cord compression, or leptomeningeal disease.
9. Patients with untreated chronic hepatitis B or HBV DNA exceeding 500IU/mL or active hepatitis C should be excluded. Patients with HCV antibody positive are eligible to participate in the study if the results of HCV RNA test show negative.
10. Known history of testing positive for human immunodeficiency virus (HIV).
11. Uncontrolled pleural effusion, pericardial effusion, or ascites requiring repeated drainage.
12. Subjects with active, known or suspected autoimmune disease, or a medical history of autoimmune disease, with the exceptions of the following: vitiligo, alopecia, Grave disease, psoriasis or eczema not requiring systemic treatment within the last 2 years, hypothyroidism (caused by autoimmune thyroiditis) only requiring steady doses of hormone replacement therapy and type I diabetes only requiring steady doses of insulin replacement therapy, or completely relieved childhood asthma that requires no intervention in adulthood, or primary diseases that will not relapse unless triggered by external factors.
13. Pregnant or lactating women.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 138 (Estimated)
Dates: Start 2021-08-23 (Actual); Primary Completion 2025-12-30 (Estimated); Study Completion 2027-01-31 (Estimated)

PRIMARY OUTCOMES:
Number of subjects experiencing dose-limiting toxicities (DLTs) | During the first 4 weeks
  DLTs will be assessed during the first 28 days of treatment and are defined as toxicities that meet pre-defined severity criteria, and assessed as having a suspected relationship to study drug, and unrelated to disease, disease progression, inter-current illness, or concomitant medications .
Adverse events (AEs) | up to 2 years
  An AE is defined as any untoward medical occurrence in a participant administered a pharmaceutical product temporally associated with the use of study treatment, whether or not considered related to the study treatment.
Objective response rate (ORR) | up to 2 years
  The ORR is defined as the proportion of subjects with CR or PR, based on RECIST Version 1.1.

SECONDARY OUTCOMES:
Progression-free survival (PFS) | Up to 2 years
  PFS is defined as the time from the date of first dosing till the first documentation of disease progression (per RECIST v1.1) or death from any cause (whichever occurs first)
Disease control rate (DCR) | Up to 2 years
  DCR is defined as the proportion of subjects with CR, PR, or SD, based on RECIST v1.1
Duration of response (DoR) | Up to 2 years
  Duration of response is defined as the duration from the first documentation of objective response to the first documented disease progression or death due to any cause, whichever occurs first.
Overall survival (OS) | up to 2 years
  OS defined as the time from the first dose to death from any cause. Subjects who do not die at the end of the extended follow-up period, or were lost to follow-up during the study, were censored at the last date they were known to be alive.
Observed pharmacokinetics (PK) exposure of AK109 and AK104 | From first dose of AK109 and AK104 through 90 days after last dose of AK109 and AK104
  The endpoints for assessment of PK of AK109 and AK104 include serum concentrations of AK109 and AK104 at different timepoints after AK109 and AK104 administration.
Number of subjects who develop detectable anti-drug antibodies (ADAs) | From first dose of AK109 and AK104 through 90 days after last dose of AK109 and AK104
  The immunogenicity of AK104 and AK109 will be assessed by summarizing the number of subjects who develop detectable anti-drug antibodies (ADAs)

CONTACTS AND LOCATIONS:
Overall Officials: Lin Shen, MD, Principal Investigator — Peking University Cancer Hospital & Institute
Locations (1):
- Beijing Cancer Hospital, Beijing, China

IPD SHARING:
Plan to Share IPD: No